CLINICAL TRIAL: NCT06167798
Title: EFFECT OF AGING ON THE GENE EXPRESSION AND HISTOMORPHOLOGY OF DENTAL GUM TISSUE
Brief Title: DENTAL GUM TISSUE AGING
Status: Completed | Type: Observational
Sponsor: The Forsyth Institute (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Sponsor
Other Study IDs: 2012007
Record Dates: First submitted 2023-12-03; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Aging
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: biopsy — two 2 mm gingival biopsies were obtained.

SUMMARY:
This is an epidemiological, cross-sectional two-visit study involving 100 Caucasian subjects representing 6 different age groups [20 to 24 (20s), 30 to 34 (30s), 40 to 44 (40s), 50 to 54 (50s), 60 to 64 (60s), and 70 to 74 (70s)]. Medically healthy subjects will receive a screening exam to determine their oral status. Subjects without periodontal disease will be enrolled in the study where two 2 mm gingival biopsy will be obtained using punch biopsy from the healthy attached gingiva around upper premolar teeth. Tissues will be processed and analyzed for histological and transcriptomics analyses targeting morphological changes and gene expression in gingival tissues with aging.

DETAILED DESCRIPTION:
This is an epidemiological, cross-sectional two-visit study involving 100 Caucasian subjects representing 6 different age groups [20 to 24 (20s), 30 to 34 (30s), 40 to 44 (40s), 50 to 54 (50s), 60 to 64 (60s), and 70 to 74 (70s)]. From each group, eighteen subjects (9 females and 9 males) will be recruited (except for the 60's and 70's groups where 14 subjects/group - 7 females and 7 males, will be recruited). At the screening visit, subjects will receive an oral soft tissue (OST) exam followed by a full periodontal exam including probing pocket depth (PPD), the difference between gingival margin and cementoenamel junction, clinical attachment level (CAL), and bleeding on probing (BOP). Subjects who meet all inclusion/exclusion criteria will receive a professional dental exam to assess the clinical status of their mouth; additionally, they will have an image of the anterior teeth taken and will fill out a questionnaire on their oral hygiene habits. At the second study visit, a 3 ml saliva sample will be collected for a saliva flow rate assessment and biomarkers analysis. Subgingival plaque samples will be taken with paper points from the tooth adjacent to the selected biopsy area, i.e. the upper second premolar. Additionally, blood (10 ml) samples for biomarker analysis and two- 2 mm-punch gingival biopsies for gene expression and histomorphology evaluations will be taken from each subject.

ELIGIBILITY:
Inclusion Criteria:

* provide written informed consent to participate in the study.
* be at the ages specified within age groups.
* male or female of the Caucasian race
* agree not to participate in any other oral/dental product studies during the course of this study.
* agree to delay any elective dentistry (including dental prophylaxis) until the study has been completed.
* agree to return for all scheduled visits and follow study procedures.
* have at least 16 natural teeth (excluding wisdom teeth).
* be in good general health, as determined by the Investigator/designee based on a review of the health history/update for participation in the study.
* healthy gingival tissue suitable for biopsy in the maxillary premolar area (per examiner discretion).

Exclusion Criteria:

* use of antibiotics 3 months prior to the study
* smoking or smoking cessation <1 year;
* any diseases or conditions to be expected to interfere with the examination or with the subject safely completing the study;
* history of drug use that is associated with gum overgrowth (i.e., dilantin, nifedipine, etc) or drugs that are known to inhibit salivary flow (i.e. antipsychotics etc.);
* chronic use of medication such as steroids, ibuprofen or acetylsalicylic acid (aspirin/ASA) more than 2-3 days/week), anti-coagulant medications, immunosuppressant medications or any other medications that in the opinion of the Investigator would interfere with the evaluation or confound interpretation of the study results. Use of low dose of ASA is permitted;
* previous gum surgery that might interfere with gum biopsy collection;
* presence or history of periodontal disease (at least 2 pockets 6mm);
* all teeth that are grossly carious, fully crowned, or extensively restored (per investigator discretion);
* any condition requiring the need for antibiotic pre-medication prior to dental procedures;
* current participation in any other oral/dental product studies;
* pregnancy or lactation;
* diabetes, autoimmune or infectious diseases, dry mouth, skin diseases;
* orthodontic appliances

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Individuals between the ages of 20-74 with healthy oral tissues will be included.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Association between age and gene expression | Through the study completion, about 6 months

IPD SHARING:
Plan to Share IPD: No